CLINICAL TRIAL: NCT00192582
Title: Relapse Prevention Trial in Top End Aboriginal People With Chronic Mental Illness
Brief Title: AIMHI NT Relapse Prevention Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menzies School of Health Research (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Alcohol Education and rehabilitation Fund (Other); Cooperative Research Centre for Aboriginal Health (Other); Northern Territory Government of Australia (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AIMHINTRPT; 283335
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychoses, Substance Induced; Depression; Bipolar Disorder
Keywords: Motivational interview; Care plan; Relapse prevention; Psychoeducation; Indigenous mental health
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Psychoses, Substance-Induced; Depression; Bipolar Disorder | interventions — Motivational Interviewing; Educational Status

INTERVENTIONS:
Behavioral: Motivational Interview with care plan and education

SUMMARY:
A new treatment for indigenous people with mental illness in remote communities has been developed. The study hypothesis is that this new treatment will result in better outcomes for clients and carers than the outcomes of clients and carers who do not receive the treatment. The treatment is a combination of a talking treatment and sharing of stories about mental health. The treatment will be delivered to the client with their chosen carer and with the local Aboriginal Mental Health Worker or Health Worker. The treatment will be given by the research team - a psychiatrist and an indigenous research officer. The trial will compare two groups of clients - a control group which is receiving 'treatment as usual', and the group which receives the new treatment. Measures of social functioning and symptoms of mental illness will be administered at base line and every six months for two years.

DETAILED DESCRIPTION:
A combined education and counselling treatment has been developed using a care plan and stories delivered via computer based animated software, with associated flip charts and information sheets. The new treatment will take about 60 minutes to administer and will be delivered on two occasions. It will include a discussion and assessment phase, setting of goals, and completion of a care plan. Three 5-minute stories will be shown during the session. Each story will have been adapted for use by the community Aboriginal Mental Health Workers prior to base line. The process for development of the stories in each community will involve showing the generic resources and any completed community specific resources - and allowing time for the stories to be adjusted by the community. The new community - specific resources will then be used in the treatment sessions - conducted by the chief investigator- a consultant psychiatrist with 15 years experience working with indigenous mental health clients and an indigenous research officer and Aboriginal Mental Health Worker (or Health Worker). The Aboriginal Mental Health Workers will receive training in the stories at two stages - through the consultation and workshop phase of the story development, and through the delivery phase with clients and carers. The stories and care planning intervention aim to promote change through encouraging clients in their own choices and their own control of their lives, and through setting goals to make changes if they choose. The intervention involves culturally appropriate sharing of information with clients and carers about illness and treatment. The information sharing is two way - as clients are invited to share their own stories during the process.

Overview

The project design is 2 years from base line to end. Base line measures of psychosocial functioning will be completed for clients and carers at commencement of the project. The measures will include self-completion and clinician completed scales. There will also be an interview - focusing on protective factors, precipitants of illness, symptoms, goals for change, and strategies for change. The new treatment will be delivered between base line and 6 weeks for group one, and in the six weeks following the six-month measures for group two. Follow up measures will be completed six months post new treatment, and every six months for 2 years post new treatment for group one. Follow up measures will be completed six months post new treatment for group two with 18 months follow up. Aboriginal Mental Health Workers will also have base line and follow up measures of knowledge and confidence in treatment - and qualitative information will be gathered about the client's progress and about the Aboriginal Mental Health Worker's experience of the new treatment.

Informed Consent

Patients, carers and Aboriginal Mental Health Workers will be given information about the project in written and spoken form, with the Aboriginal research officer, prior to obtaining their consent to participate.

Recruitment of participants Participants will be recruited by Aboriginal Mental Health Workers - or nominated by mental health staff or the General Practitioner. The treating doctors will be notified of the nomination in each case and, if they have no concerns, the Aboriginal Mental Health Worker will arrange the information and consent session with the research team. The participants will be clients who have a primary chronic mental illness, are aged over 18 years, are able to give informed consent, and are current clients. The diagnoses for inclusion are Schizophrenia, Delusional disorder, Schizoaffective disorder, Drug-induced psychosis, Non-specific psychoses, and Affective psychoses. People with Intellectual disability or organic brain disorders will be excluded. The criteria for chronicity for the purposes of the project are defined by two or more episodes of illness severe enough to require medical intervention and treatment. The carer will be identified by discussion between the client and the Aboriginal Mental Health Worker or Health Worker.

Random allocation to two groups within communities The consenting clients and carers will be allocated within communities randomly to Group 1 (treatment group) and Group 2 (control group). The researchers will not direct the allocation or be involved in choosing the groups. The control group will still receive the new treatment - but they will receive the new treatment 6 months after Group 1.

Baseline measures

Baseline data will be collected on all consumers at base line - gender, age, place of residence, psychiatric and alcohol and other drug history, social history, family situation, strengths and skills. The number of people in the home and home stressors will also be recorded. A formal psychiatric diagnosis will be applied following review of history and previous diagnoses, and base line measures. Measures will be taken at base line and every six months up to 2 years. The new treatment will be given twice - once after the base line measures are completed and a follow up session 2 to 6 weeks later. The measures rate symptoms, social functioning. substance dependence and the client's knowledge of their illness. The following three brief base line and follow up measures will be used for clients in addition to the interview.

Client rated scales

Partners in Health Scale (PIH), Kessler 10, Severity of Dependence Scale,

Carer rated scales

The carer will be interviewed with the client. There will be two occasions when the carer is asked for a separate rating - their own K10 and their view of the client's substance misuse worry score.

Clinician rated scales Health of the Nation Outcome Scales, Life Skills Profile, Global Assessment of Functioning,

Clinical File Audit

A file audit at base line and at 12 months and 2 years will score the following:

Mental health assessment recorded in preceding 3 months Involvement of specialist mental health services in assessment and treatment planning Early warning signs recorded Causes of getting sick again noted Strategies to address causes of getting sick again incorporated in treatment plan Care Plan developed Care Plan goals reviewed Service contact, hospital admission, number of hospital days, and mental health act detention data will also be reviewed. This routinely collected data will be examined by the research team for number of attendances of the client at the health clinic, service events by the regional mental health service, and hospital admission and detention occasions in the 12 months prior to the project and for the 2 years duration of the project.

Interview - Qualitative data

A clinical assessment and a care plan will be completed. There will be a semi-structured discussion about the client's experience of mental illness, which will be recorded by written notes. The AMHW, carer, and indigenous research officer will be present. At any time the carer will only be present if the client gives consent to that. This interview will cover symptoms, treatment, and goals for change, barriers to change, and strategies for change. After the second new treatment the client and carer will be asked their opinion of the care package and whether they found it easy to use, interesting and acceptable, and whether they believed it had changed their knowledge or attitudes to illness in any way and if so - in what way.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited by Aboriginal Mental Health Workers - or nominated by mental health staff or the General Practitioner. The treating doctors or local mental health team will be notified of the nomination in each case and, if they have no concerns, the Aboriginal Mental Health Worker will arrange the information and consent session with the research team. The participants will be clients who have a primary chronic mental illness, are aged over 18 years, are able to give informed consent, and are current clients. The diagnoses for inclusion are Schizophrenia, Delusional disorder, Schizoaffective disorder, Drug-induced psychosis, Non-specific psychoses, and Affective disorders. The criteria for chronicity for the purposes of the project are defined by two or more episodes of illness severe enough to require medical intervention and treatment. The carer will be identified by discussion between the client and the Aboriginal Mental Health Worker or Health Worker.

Exclusion Criteria:

People aged less than 18 years, and people with known Intellectual disability or organic brain disorders will be excluded. People with illnesses which have not recurred, or which are not likely to recur will be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2005-07; Study Completion 2007-08 (Estimated)

PRIMARY OUTCOMES:
Health of Nations Outcome Scale (HONOS) | Baseline, 6 months, 12 months, 18 months,

SECONDARY OUTCOMES:
Life Skills Profile 16 (LSP) | Baseline, 6 months, 12 months, 18 months,
Severity of Dependence Scale (SDS) | Baseline, 6 months, 12 months, 18 months,
Kessler 10 - client and carer | Baseline, 6 months, 12 months, 18 months,
Partners in Health Scale (PIH) - modified | Baseline, 6 months, 12 months, 18 months,
Semi structured interview with carer and client and Aboriginal Mental Health Worker | Baseline, 6 months, 12 months, 18 months,

CONTACTS AND LOCATIONS:
Overall Officials: Tricia M Nagel, MBBS, FRANZCP, Principal Investigator — Menzies School of Health Research, Australia
Locations (1):
- Menzies School of Health Research, Darwin, Northern Territory, Australia

REFERENCES:
- [Derived] Nagel T, Robinson G, Condon J, Trauer T. Approach to treatment of mental illness and substance dependence in remote Indigenous communities: results of a mixed methods study. Aust J Rural Health. 2009 Aug;17(4):174-82. doi: 10.1111/j.1440-1584.2009.01060.x. PMID 19664081